CLINICAL TRIAL: NCT04475627
Title: Inter-field Strength Agreement of Myocardial Strain Measurements Using Cardiovascular Magnetic Resonance Imaging
Brief Title: Inter-field Strength Agreement of CMR Derived Strain
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0735
Record Dates: First submitted 2020-07-02; First posted 2020-07-17 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular magnetic resonance; left ventricular strain; field strength
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants randomised to 1.5T then 3T: Participants randomized to be scanned at 1.5T first followed by 3T
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) imaging at 1.5T; Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) imaging at 3T
- Participants randomised to 3T then 1.5T: Participants randomized to be scanned at 3T first followed by 1.5T
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) imaging at 1.5T; Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) imaging at 3T

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) imaging at 1.5T — Long and short axis bSSFP cines images, long and short axis tagging images and aortic cine images will be obtained. Participants will be randomised to either have cine or tagging images obtained first.
Diagnostic Test: Cardiovascular Magnetic Resonance (CMR) imaging at 3T — Long and short axis bSSFP cines images, long and short axis tagging images and aortic cine images will be obtained. Participants will be randomised to either have cine or tagging images obtained first.

SUMMARY:
* Magnetic Resonance Imaging (MRI) scanners create a strong magnetic field around the body to produce a detailed picture of parts of the body. This can provide a lot of useful information about how the heart looks and works.
* Different strengths of magnets can be used in an MRI scanner and this can affect the pictures that are produced. To scan the heart, two different magnet field strengths (1.5 tesla (T) and 3T) are mainly used.
* It is currently unclear if when the heart is scanned using these different field strengths, if the measurements that tell us how well the heart squeezes and relaxes (known as 'myocardial strain') will be the same between them.
* This study is investigating if myocardial strain measurements using 1.5T and 3T MRI scanners are different or if they can be used interchangeably.
* Twenty healthy people without heart disease will be recruited to have two MRI scans on the same day. The order that they have their scan (either on a 1.5T MRI scanner first or a 3T MRI scanner first) will be decided randomly.
* All images will then be analysed using specialist software to provide measurements of myocardial strain. These measured can then assessed to see if there is agreement between the myocardial strain results at the two MRI field strengths.

DETAILED DESCRIPTION:
* This is a single-centre, randomised, cross-sectional, cross-over observational study.
* Twenty healthy volunteers, aged 18 years and over will be recruited and will undergo cardiovascular magnetic resonance scans for long axis and short axis cine imaging at 1.5T and 3T.
* Participation will involve one single visit where participants will be consented, randomised and then undergo scanning at both field strengths; the order of scanning at 1.5T and 3T will be randomised. There will be no follow up period.
* All subjects will undergo balanced steady-state free precession (bSSFP) cine imaging at 3T and 1.5T. Tagging images will also be acquired at both field strengths. Participants will also be randomized to either have cine or tagging images obtained first on each scan.
* All scans at both field strengths will be anonymised and analysed offline by a single experienced observer to determine inter-field strength agreement of left ventricular systolic and diastolic strain measurements.
* Further imaging analysis will take place for secondary outcomes, including analysis using other software vendors, tagging images and aortic cine images.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Understands written and verbal English sufficiently to be able to consent and participate in study
* Male or Female, aged 18 years or above.
* No history of cardiovascular, respiratory, metabolic (including diabetes) or renal disease.

Exclusion Criteria:

* Prior cardiovascular, respiratory, metabolic (including diabetes) or renal disease.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Any contra-indication to magnetic resonance imaging (MRI), including the presence of an implanted metal device or suspected metal foreign bodies.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, male and female, aged 18 years or above
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Inter-field strength agreement of left ventricular global longitudinal strain (GLS) | Day 1
  The inter-field strength agreement of left ventricular global longitudinal strain (GLS) measured using cvi42 Tissue Tracking at 1.5T and 3T

SECONDARY OUTCOMES:
Inter-field strength agreement of left ventricular global circumferential strain (GCS) | Day 1
  The inter-field strength agreement of left ventricular global circumferential strain (GCS) measured using cvi42 Tissue Tracking at 1.5T and 3T
Inter-field strength agreement of left ventricular short- and long-axis global radial strain (GRS) | Day 1
  The inter-field strength agreement of left ventricular short- and long-axis global radial strain (GRS) measured using cvi42 Tissue Tracking at 1.5T and 3T
Inter-field strength agreement of left ventricular longitudinal peak early diastolic strain rate (long. PEDSR) | Day 1
  The inter-field strength agreement of left ventricular longitudinal peak early diastolic strain rate (long. PEDSR) measured using cvi42 Tissue Tracking at 1.5T and 3T
Inter-field strength agreement of left ventricular circumferential peak early diastolic strain rate (circum. PEDSR) | Day 1
  The inter-field strength agreement of left ventricular circumferential peak early diastolic strain rate (circum. PEDSR) measured using cvi42 Tissue Tracking at 1.5T and 3T
Inter-field strength agreement of left ventricular radial peak early diastolic strain rate (rad. PEDSR) | Day 1
  The inter-field strength agreement of left ventricular radial peak early diastolic strain rate (rad. PEDSR) measured using cvi42 Tissue Tracking at 1.5T and 3T
Inter-field strength agreement of left ventricular peak torsion | Day 1
  The inter-field strength agreement of left ventricular peak torsion measured using cvi42 Tissue Tracking at 1.5T and 3T
Inter-vendor agreement of left ventricular systolic and diastolic strain measurements at 1.5T and 3T | Day 1
  The inter-vendor agreement of left ventricular systolic and diastolic strain measurements with different software packages (TomTec, QMass, cvi42) using cine-based imaging at 1.5T and 3T
Inter-field strength agreement of left ventricular systolic and diastolic strain measurements using cine-based imaging and tissue tagging techniques | Day 1
  The inter-field strength agreement of left ventricular systolic and diastolic strain measurements derived using cine-based imaging and tissue tagging techniques at 1.5T and 3T
Inter-field strength agreement of left and right atrial and ventricular volumes and function | Day 1
  The inter-field strength agreement of left and right atrial and ventricular volumes and function at 1.5T and 3T
Inter- and intra-observer variability of left ventricular systolic and diastolic strain measurements | Day 1
  The inter- and intra-observer variability of left ventricular systolic and diastolic strain measurements using cvi42 Tissue Tracking at 1.5T and 3T
Inter-field strength agreement of aortic strain | Day 1
  The inter-field strength agreement of aortic strain measured at 1.5T and 3T

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No